CLINICAL TRIAL: NCT00542360
Title: Marketing Fall Prevention Classes to Older Adults in Faith-Based Congregations: Cluster Randomized Controlled Trial
Brief Title: Marketing Fall Prevention Classes to Older Adults in Faith-Based Congregations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Colorado State University (Other); Colorado Department of Public Health and Environment (Other Government); University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 06-0636
Record Dates: First submitted 2007-10-09; First posted 2007-10-11 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Accidental Falls
Keywords: Accidental Falls; Aged; Social Marketing; Exercise; Accident Prevention; Religion; Randomized Controlled Trial
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Social marketing program (Experimental): Behavioral: Social marketing program to motivate exercise class participation
  Interventions: Behavioral: Marketing program to motivate exercise class participation
- Control (No Intervention): Control: No intervention

INTERVENTIONS:
Behavioral: Marketing program to motivate exercise class participation — Using qualitative research methods, a targeted social marketing program, including a 'marketing toolkit,' was developed to motivate participation in exercise classes by older adult members of churches. The Health Belief and Transtheoretical Models formed the theoretical basis for the social marketing planning process and guided program design. The marketing program aimed to increase exercise class attractiveness, usability, and uptake by reducing barriers and costs, and using messaging about benefits and enhanced convenience to motivate participation. The intervention was implemented through churches.
  Arms: Social marketing program

SUMMARY:
This cluster randomized trial will test whether a social marketing program implemented in churches can motivate older adults to join exercise classes, in order to improve their strength and balance and thus prevent falls.

DETAILED DESCRIPTION:
Injuries from falls are a leading cause of emergency visits, hospitalizations, and deaths in older US adults, resulting in total lifetime costs of more than $19 billion in 2000. Fall injuries reduce independence and mobility, and increase disability and institutionalization. There is good evidence that community-based group exercise classes focusing on strength and balance prevent older adult falls, but uptake is limited. This study will test a new approach to promote participation in group balance-retraining exercise classes, targeting older adults in faith-based congregations. The proposal addresses national research priorities to evaluate strategies for dissemination and implementation of effective interventions to prevent falls among community-dwelling older adults. Focus groups and key informant interviews will provide research-based understanding of church members aged 60+ and those who influence them, and explore facilitators and barriers to class participation. With this formative research, a targeted social marketing program will be developed to motivate participation. Behavioral change and social marketing theories form the intervention's theoretical basis and will guide program design. The marketing program aims to increase class attractiveness, usability, and uptake by reducing barriers or costs and using incentives or other benefits to reinforce participation. Churches, representing varied denominations and communities, will be randomly allocated to intervention (marketing program implementation) or control (no program) groups. Outreach to diverse churches will ensure that materials and strategies target potentially hard-to-reach (e.g., Hispanic, rural) populations. The trial will test whether older adult members of intervention churches are more likely to join balance retraining classes. Factors that may mediate intervention effects will be examined. Secondary outcomes include baseline fall risk among class participants, assessed by physical function tests; and intensity, diffusion, message penetration and acceptability of the marketing program, and persistent facilitators and barriers to class participation, evaluated with process measures, focus groups, and structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* Churches located in Mesa County, Colorado, that have adult members who are aged 60 and older
* Exercise class participants will include community-dwelling members of enrolled churches who are aged 60 and older, English- or Spanish-speaking, ambulatory with or without assistive devices, and cognitively able to consent and be tested.

Exclusion Criteria:

* Older adults with any medical condition that precludes participation in an exercise program, as determined by the participant or their physician, or who are not physically able to pass the Modified-Clinical Test of Sensory Interaction in Balance (M-CTSIB) at baseline

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-10; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is defined as attending at least one balance-retraining exercise class designed to reduce older adult falls | During the two-year intervention period

SECONDARY OUTCOMES:
Baseline fall-risk status of participants who attend at least one balance-retraining exercise class for fall prevention | During the two-year intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn G DiGuiseppi, MD, MPH, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Colorado Department of Public Health and Environment, Grand Junction, Colorado

REFERENCES:
- [Background] Clark L, Thoreson S, Goss CW, Zimmer LM, Marosits M, DiGuiseppi C. Understanding fall meaning and context in marketing balance classes to older adults. J Appl Gerontol. 2013 Feb;32(1):96-119. doi: 10.1177/0733464811399896. Epub 2011 Apr 1. PMID 25473927
- [Background] Currie DW, Thoreson SR, Clark L, Goss CW, Marosits MJ, DiGuiseppi CG. Factors Associated With Older Adults' Enrollment in Balance Classes to Prevent Falls: Case-Control Study. J Appl Gerontol. 2020 Aug;39(8):908-914. doi: 10.1177/0733464818813022. Epub 2018 Nov 18. PMID 30451055
- [Result] DiGuiseppi CG, Thoreson SR, Clark L, Goss CW, Marosits MJ, Currie DW, Lezotte DC. Church-based social marketing to motivate older adults to take balance classes for fall prevention: cluster randomized controlled trial. Prev Med. 2014 Oct;67:75-81. doi: 10.1016/j.ypmed.2014.07.004. Epub 2014 Jul 12. PMID 25025522
- [Derived] Clark L, Thoreson S, Goss CW, Marosits M, Zimmer LM, Flattes V, DiGuiseppi C. Older Adults' Perceptions of a Church-Based Social Marketing Initiative to Prevent Falls Through Balance and Strength Classes. J Appl Gerontol. 2021 Nov;40(11):1475-1482. doi: 10.1177/0733464820984288. Epub 2021 Jan 6. PMID 33406989